CLINICAL TRIAL: NCT06418984
Title: A Randomized Clinical Trial to Compare the Influence of Optimized Attachments, IPR and a Combination of Both Techniques on the Rotational Accuracy of Canines With Clear Aligners
Brief Title: Clinical Trial to Compare Clear Aligners' Auxiliaries on Rotational Accuracy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202400491
Record Dates: First submitted 2024-05-08; First posted 2024-05-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-03

CONDITIONS: Rotation of Tooth

STUDY DESIGN:
Intervention Model Description: one control group and 3 experimental groups
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Control (No Intervention): No Interproximal reduction or attachments will be used to help correct the rotation
- Inter proximal reduction (Experimental): Interproximal reduction will be performed in this arm
  Interventions: Device: auxiliary
- Optimized attachments (Experimental): optimized composite attachments will be added to this arm
  Interventions: Device: auxiliary
- IPR and optimized attachments (Experimental): Both Interproximal reduction will be implemented and optimized attachments will be added to this arm
  Interventions: Device: auxiliary

INTERVENTIONS:
Device: auxiliary — the interventions are related to the adjuncts associated with clear aligners to improve the predictability and accuracy of tooth movement
  Arms: IPR and optimized attachments; Inter proximal reduction; Optimized attachments

SUMMARY:
This randomized clinical trial aims to assess the effectiveness of optimized attachments, IPR and a combination of the two techniques on the rotational accuracy of canines with clear aligners

DETAILED DESCRIPTION:
Study Visit 1 (V1): Upon fitting the inclusion criteria, the patient will be randomized to one of the four interventional groups. A member of the study team will collect the initial orthodontics records. These records include two radiographs (a panoramic radiograph and a lateral cephalogram), intraoral and extraoral photographs, and an iTero intraoral digital scan. The scan will be sent directly to the Align Technology Invisalign doctor platform to begin the process of fabricating the desired aligners according to the clinical instructions for the simulated treatment plan by the study team and the randomly assigned group for the patient. Study Visit 2 (V2): 5 weeks following visit 1, Invisalign aligners will be delivered to the included and randomized subjects, and associated treatment rendered. Subjects will be instructed to wear their aligners full-time except while eating, drinking, and brushing and change their aligners as recommended by Invisalign® every week. Study Visit 3 (V3): The trial will end after the patient has completed wearing the first stage of aligners. Final records will be collected: these include iTero intraoral digital scans to construct the 3D digital models, intraoral and extraoral photographs, and radiographs.

To assess the accuracy of the achieved outcomes and compare the outcomes of the four treatment groups, the collected digital models (predicted simulated models and achieved final scanned models) will be superimposed and compared to assess the accuracy and predictability of rotational tooth movement in the included subjects, and treatment outcomes will be evaluated. The differences between the positions of each tooth in the two digital models (predicted from Clincheck and achieved from the final scan) will quantified for rotation: differences of 2° or more rotation will be considered clinically relevant. These values were chosen from the American Board of Orthodontics (ABO) model grading system for case evaluation and other clinical studies.5 Additionally, data related to treatment duration, number of aligners, and number of visits needed to complete the treatment will be gathered and analyzed in a de-identified form.

ELIGIBILITY:
Inclusion Criteria

* Physically healthy with no relevant allergies or medical problems
* Male or female above 18 years old
* Full permanent dentition except for the third molars
* Any type of malocclusion with rotated canines that require derotation
* Good oral hygiene and absence of periodontal disease
* Malocclusion to be treated with Invisalign aligners (SmartTrack)
* Any ethnic group

Exclusion Criteria

* Orthognathic surgical cases
* An extraction treatment plan
* Poor oral hygiene
* Patients with syndromes or craniofacial anomalies.
* The use of any other orthodontic appliance than clear aligners' (Invisalign)
* Malocclusion that requires auxiliaries in the simulated plan ( buttons and elastics on the canines)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-28 (Actual)

PRIMARY OUTCOMES:
Accuracy of Canine rotation | 6-9 months
  3D model superimposition will be used to assess the accuracy of tooth movement

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States